CLINICAL TRIAL: NCT00321516
Title: Effects of Aripiprazole on the Steady-State Pharmacokinetics of Lamotrigine in Subjects With Bipolar I Disorder
Brief Title: Drug-drug Interaction Study of Aripiprazole and Lamotrigine in Patients With Bipolar Type I Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CN138-402; IND #: 42,776
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2008-06

CONDITIONS: Bipolar Disorder
Keywords: Bipolar type I Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: aripiprazole

INTERVENTIONS:
Drug: aripiprazole — Tablets, Oral, 10, 20, or 30 mg (titrated), once daily, 14 days.
  Other Names: Abilify

SUMMARY:
The purpose of this clinical research study is to learn if aripiprazole has a drug-drug interaction with lamotrigine.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18 to 40 kg/m2
* Subjects with bipolar I disorder who are clinically stable on a stable dose of at least 100 mg lamotrigine for at least 4 weeks prior to study entry
* Men and women, ages 18 to 65

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Patients with any significant acute or chronic medical illness, other than bipolar I disorder
* Subjects with active psychotic symptoms
* History of head trauma within the past 2 years
* History of akathisia requiring treatment
* History of tardive dyskinesia or abnormal involuntary movements
* Subjects with a predisposition to orthostatic hypotension
* Positive urine screen for drugs of abuse
* Use of narcotic-containing agents, amphetamines, or hormonal contraceptives within 4 weeks of study start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Comparison of Cmax (maximum drug concentration) and AUC(Tau) (exposure) of lamotrigine at the beginning of the study (Day-1) and when the subject completes the study (Day 36)

SECONDARY OUTCOMES:
Assess the safety and tolerability of aripiprazole when co-administered with lamotrigine for up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Austin, Texas
  - Local Institution, Bellaire, Texas
  - Local Institution, Desota, Texas